CLINICAL TRIAL: NCT06088966
Title: Evaluation of Hemodynamic and Ventilatory Effects of Negative Pressure Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karlsburg Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Matthias Heringlake, Clinical Professor and head of the department of anesthesiology and intensive care Prof. Dr. Matthias Heringlake, Karlsburg Hospital
Other Study IDs: KAIKB-2023-2
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigation of the effects of negative pressure ventilation after cardiac surgery in adults onto performance of the left and right heart and the lungs.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary artery catheter after cardiac surgery

Exclusion Criteria:

* minimally invasive surgery
* unstable conditions
* bleeding
* unability to fit cuirass

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients after surgery without exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Stroke Volume Index in ml/m2 | 1 hour

SECONDARY OUTCOMES:
Heart rate in beats/min | 1 hour
blood pressure in mm/Hg | 1 hour
arterial oxygen saturation in % | 1 hour
mixed venous oxygen saturation in % | 1 hour
  measured via pulmonary catheter
right ventricular ejection fraction in % | 1 hour
  measured via pulmonary catheter
end diastolic volume index in ml/m2 | 1 hour
  measured via pulmonary catheter
Cardiac index in l/min/m2 | 1 hour
  measured via pulmonary catheter
tricuspid annular plane systolic excursion in mm | 1 hour
  measured via transesophageal echocardiography
right ventricular fractional area change in % | 1 hour
  measured via transesophageal echocardiography
Vena contract of tricuspid valve in mm | 1 hour
  measured via transesophageal echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Karlsburg, Klinik für Anästhesiologie, Karlsburg, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Schemke S, Grunewald H, Schemke L, Franzen K, Hirschl D, Heringlake M, Muras L. A pilot study on the hemodynamic effects of negative pressure ventilation in patients after cardiac surgery focussing on right ventricular function. Sci Rep. 2025 Jul 31;15(1):27974. doi: 10.1038/s41598-025-12534-1. PMID 40744972